CLINICAL TRIAL: NCT00407693
Title: PET Whole Body Imaging Using a Peripheral Benzodiazepine Receptor Ligand [C-11]PBR28
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 070035; 07-M-0035
Record Dates: First submitted 2006-12-02; First posted 2006-12-05 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2016-07-21

CONDITIONS: Healthy
Keywords: Dosimetry; Effective Dose; Radiation-Absorbed Dose

INTERVENTIONS:
Drug: [C-11]PRB28

SUMMARY:
In this study we will examine where the radioactive tracer [11C]PBR28 is distributed in the body of healthy volunteers to calculate the radiation exposure to organs of the body. We will also test if [11C]PBR28 binds to your blood cells and compare with the binding in PET images.

DETAILED DESCRIPTION:
The peripheral benzodiazepine receptor (PBR) is distinct from central benzodiazepine receptors associated with GABA(A) receptors. Although PBR was initially identified in peripheral organs such as kidneys, endocrine glands and lungs, later studies identified PBR in the central nervous system. In normal conditions, PBR is expressed in low levels in some neurons and glial cells. PBR can be a clinically useful marker to detect neuroinflammation because activated microglial cells in inflammatory areas express much greater levels of PBR than in microglial cells in resting conditions.

PBR has been imaged with positron emission tomography (PET) using [(11)C]1-(2-chlorophenyl-N-methylpropyl)-3-isoquinoline carboxamide (PK11195). However, this classical ligand provides only low levels of specific signals and is not sensitive to detect changes that occurred in vivo. Recently we developed a new ligand, N-acetyl-N-(2-[(11)C]methoxybenzyl)-2-phenoxy-5-pyridinamine [(11)C]PBR28), which showed much greater specific signals than [(11)C]PK11195 in non-human primates. Therefore, [(11)C]PBR28 is a promising PET ligand. However, radiation absorbed doses have not been estimated from human whole body imaging.

The initial purpose of this protocol is to estimate radiation absorbed doses of [11C]PBR28 by performing whole body imaging studies on ten healthy human subjects. The radiation absorbed doses are required to apply this PET ligand in various neurological and psychiatric disorders in the future.

Under the current and other protocols using [(11)C]PBR28, we found that some healthy subjects and patients have very low to no binding of [(11)C]PBR28. We studied approximately 188 subjects in total under protocols using [11C]PBR28 and found that 8.5% (16/188) had almost no binding of [(11)C]PBR28. Several published ligands have been tested and all of the tested ligands recently developed show low affinity to a subset of humans. By using [(11)C]PBR28, we need to exclude PBR28 nonbinders from the data to study changes in PBR. By using a PET ligand that binds equally to PBR28 binders and nonbinders, we would be able to study all subjects. We also confirmed that PBR28 nonbinders determined by PET do not show binding in in vitro binding assays using blood cells.

We wish to test new ligands currently being developed in our chemistry group by obtaining blood samples from additional PBR28 nonbinders (= low affinity binders) and by performing in vitro binding assays. Because our preliminary analysis of whole body imaging has shown that the differences between PBR28 binders and nonbinders might somewhat vary among organs and the cause of the nonbinding phenomenon is not fully understood, after identifying PBR28 nonbinders by binding assays, we will perform whole body imaging using [(11)C]PBR28.

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects must be healthy and aged 18-65 years.

EXCLUSION CRITERIA:

* Current psychiatric disease, substance abuse or severe systemic disease based on history and physical exam.
* Laboratory tests with clinically significant abnormalities.
* Prior participation in other research protocols or clinical care in the last year such that radiation exposure including that from this protocol would exceed the guidelines set by the Radiation Safety Committee (RSC).
* Pregnancy and breast feeding.
* Positive HIV test.
* Cannot lie flat for 2 - 3 h.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-11-28; Study Completion 2016-07-21 (Actual)

PRIMARY OUTCOMES:
Biodistribution of [C-11]PBR28

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Fujita, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anholt RR, De Souza EB, Oster-Granite ML, Snyder SH. Peripheral-type benzodiazepine receptors: autoradiographic localization in whole-body sections of neonatal rats. J Pharmacol Exp Ther. 1985 May;233(2):517-26. PMID 2987488
- [Background] Anholt RR, Murphy KM, Mack GE, Snyder SH. Peripheral-type benzodiazepine receptors in the central nervous system: localization to olfactory nerves. J Neurosci. 1984 Feb;4(2):593-603. doi: 10.1523/JNEUROSCI.04-02-00593.1984. PMID 6321699
- [Background] Anholt RR, Pedersen PL, De Souza EB, Snyder SH. The peripheral-type benzodiazepine receptor. Localization to the mitochondrial outer membrane. J Biol Chem. 1986 Jan 15;261(2):576-83. PMID 3001071